CLINICAL TRIAL: NCT01230242
Title: Experimental Study Examining Mirena IUD Insertion and Estimating Rates of Expulsion Immediately After Placental Delivery.
Brief Title: Postplacental Mirena IUD Insertion and Estimating Expulsion Rates.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended to determine if Mirena device could be charged to patient insurance
Sponsor: Rebecca Hunt (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor-Investigator, Rebecca Hunt, Physician, MMP Women's Health Maternal-Fetal Medicine, MaineHealth
Organization: MaineHealth (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3689
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Results first posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Estimating Rates of Expulsion
Keywords: Mirena; postplacental intrauterine device; postpartum insertion

STUDY DESIGN:
Intervention Model Description: Mirena IUD placement
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mirena IUD Placement Immediately Post-delivery (Experimental): Participants enrolling in this study agree to have the IUD placed immediately post-delivery versus waiting the standard 6 weeks.
  Interventions: Device: Levonorgestrel Intrauterine Device

INTERVENTIONS:
Device: Levonorgestrel Intrauterine Device — levonorgestrel intrauterine device insertion within ten minutes of placental delivery using a ring forceps insertion protocol
  Other Names: Mirena

SUMMARY:
This study aims to demonstrate that the expulsion rate is increased but acceptable when inserting Mirena IUDs immediately postpartum, termed 'postplacental IUD insertion'. The investigators will compare the postplacental insertion expulsion rate estimate with rates reported in the literature for 6 week postpartum insertion, which is currently the American standard for IUD insertion postpartum. Secondary outcomes will also be examined; endometritis, uterine perforation, continuation and pregnancy among others.

DETAILED DESCRIPTION:
The average expulsion rate for 6 week postpartum IUD insertion is approximately 10-12% with a range between 3-20% at 1 year. An acceptable expulsion rate for postplacental insertion (PPI) has not been defined and varies between studies. There are limited data on the expulsion rates of levonorgestrel intrauterine systems. Expulsion rates range widely from 1-3% to as high as 30-40% depending on the IUD and the study. Studies report an average rate of expulsion in ranges approximating 10-12%, similar to 6 week insertion rates.

There are many limitations to published studies including the use of older model IUDs no longer in use, multiple insertion techniques that have been deemed ineffective in reducing expulsion rates as well as varying follow up times making comparison of expulsion rates difficult.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or greater
* obstetric patient in greater Portland, ME area

Exclusion Criteria:

* Evidence of chorioamnionitis (persistent fetal tachycardia, intra-partum fever >38.0)
* prolonged rupture of membranes (greater than 24 hours)
* intrauterine fetal demise
* use of general anesthesia at time of delivery
* postpartum hemorrhage (>500ml vaginal, >1000ml cesarean)
* magnesium administration in labor due to HELLP syndrome or preeclampsia
* preterm delivery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-09-07 (Actual); Primary Completion 2010-10-27 (Actual); Study Completion 2011-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Mueller, MD, Principal Investigator — MaineHealth

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 4 subjects were consented out of the 20. Of those 4 only 3 had the IUD inserted.
Groups:
- Mirena IUD Placement Immediately Post-delivery: Subjects to have Mirena IUD Placement Immediately Post-delivery
Period: Overall Study
Arm/Group | Mirena IUD Placement Immediately Post-delivery
Started | 4
Completed | 1
Not Completed | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mirena IUD Placement Immediately Post-delivery
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Expelled IUDs by12 Weeks Postpartum
Description: Number of participants who expelled IUDs by12 weeks postpartum across all participants
Time Frame: up to 12 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Mirena IUD Placement Immediately Post-delivery
Number analyzed (Participants) | 4
Participants | 1

ADVERSE EVENTS:
Time Frame: 12 weeks post IUD placement
Arm/Group | Mirena IUD Placement Immediately Post-delivery
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes